CLINICAL TRIAL: NCT05035836
Title: A Phase 2 Single-Arm Open-Label Pilot Trial Evaluating Zanidatamab (ZW25) in Patients With Early Stage HER2/Neu Positive (HER2+) Breast Cancer (BC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Zymeworks BC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0358; NCI-2021-09420 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; HER2-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — zanidatamab; Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zanidatamab (Experimental): zanidatamab by vein every 2 weeks (+/- 3 days) for up to 6 doses (3 study cycles
  Interventions: Drug: Zanidatamab; Drug: Letrozole; Drug: Tamoxifen

INTERVENTIONS:
Drug: Zanidatamab — Given IV
  Other Names: ZW25
Drug: Letrozole — Given by PO
Drug: Tamoxifen — Given by PO

SUMMARY:
This is a Phase 2, single-site, single-arm open-label trial of zanidatamab in patients with early stage, low risk HER2+ BC.

The primary objective is to determine the efficacy of zanidatamab for patients with early stage HER2/neu positive (HER2+) breast cancer (BC) as determined by pathologic complete response (pCR) .

DETAILED DESCRIPTION:
Primary Objective:

To determine the efficacy of zanidatamab for patients with early stage HER2/neu positive (HER2+) breast cancer (BC) as determined by pathologic complete response (pCR) 1

Secondary Objective(s):

* To determine pathologic response by residual cancer burden (RCB). 1-3
* To evaluate the radiographic response and volumetric change in tumor size by ultrasound and MRI
* To evaluate tolerability and safety of zanidatamab for treatment-naïve early stage HER2+ breast cancer (BC).
* To evaluate the rate of adverse events and treatment-emergent adverse events with zanidatamab alone (for patients with hormone receptor negative tumors) or with endocrine therapy tamoxifen or letrozole (in hormone receptor positive tumors)
* To evaluate the feasibility of treating patients with early stage HER2+ breast cancer with monotherapy zanidatamab
* To determine tumor-based predictive biomarkers of response

Exploratory Objective(s):

* To assess circulating free DNA levels and dynamics as biomarkers of response
* To assess effect of zanidatamab on immune environment

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give written informed consent
2. Age > 18 years at time of study entry.
3. Patient would be willing to undergo surgery is appropriate for surgery
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 1).
5. Tumor size > 1 cm to ≤ 3 cm assessed by ultrasound and clinically and radiographically node negative with no known metastatic disease.
6. HER2+ BC as defined by American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) guidelines.31 Patients may have ER+ or ER- negative disease, as defined by ASCO-CAP guidelines.
7. Left ventricular ejection fraction (LVEF) must be within institutional limits of normal as assessed by echocardiogram (ECHO) or multigated acquisition (MUGA) scan, documented within 4 weeks prior to first dose of study drug.
8. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (≥ 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (≥100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). The maximum allowable bilirubin is ≤ 2.5 x ULN for patients with Gilbert's disease.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional ULN
   * Calculated glomerular filtration rate >50 mL/min
9. Patients must either be of non-reproductive potential or willing to undergo appropriate contraception. Male subjects must agree not to donate sperm and female subjects must agree not to donate oocytes starting at screening and throughout the study period, and for at least 12 months after treatment discontinuation.
10. Patient with reproductive potential must have a negative pregnancy test ≤3 days prior to the first dose of zanidatamab.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Involvement in the planning and/or conduct of the study.
2. Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
3. Has received therapy for this current diagnosis of BC including investigational therapy, endocrine therapy, targeted therapy, or chemotherapy, surgery or radiation.
4. Mean QT interval corrected for heart rate (QTc) ≥ 470 ms.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active peptic ulcer disease or gastritis, active bleeding diatheses, , or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent.
6. Female patients who are pregnant, breast-feeding, or of reproductive potential who are not employing an effective method of birth control.
7. Patients with uncontrolled seizures.
8. Any major surgery for any reason, within 4 weeks of the enrollment. Portacath placement will be allowed.
9. Clinically significant cardiac disease such as ventricular arrhythmia requiring therapy, , myocardial infarction, unstable angina (within 6 months prior to first dose of study drug), any history of cardiac failure, and uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
10. Known active Hepatitis B and/or Hepatitis C. Hepatitis testing is not required unless the patient has a history of Hepatitis B or C.
11. Known to be HIV positive. HIV testing is not required for those patients who are not known to be positive.
12. Total lifetime anthracycline load exceeding 360 mg/m2 doxorubicin or equivalent
13. Any condition that requires systemic treatment with either corticosteroids (>10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤14 days prior to randomization. Note: Subjects who are currently or have previously been on any of the following steroid regimens are not excluded:

    1. Adrenal replacement steroid (dose ≤10 mg daily of prednisone or equivalent)
    2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption\
    3. Short course (≤7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
14. History of life-threatening hypersensitivity to monoclonal antibodies or to recombinant proteins or excipients in the drug formulation
15. Known distant metastatic disease including (CNS) metastases, symptomatic CNS metastases, and leptomeningeal disease (LMD).
16. Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease (with exception of subjects with Gilbert's Syndrome, asymptomatic gall stones, liver metastases, or stable chronic liver disease per investigator assessment)
17. Symptomatic pulmonary embolism ≤28 days
18. Administered a live vaccine ≤4 weeks prior to randomization. Patients can get COVID vaccine that are not alive before ot during the study period, with 48 hours between vaccine administration and investigation agent administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2028-12-29 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of zanidatamab for patients with early stage HER2/neu positive (HER2+) breast cancer (BC) as determined by pathologic complete response (pCR | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vicente Valero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org